CLINICAL TRIAL: NCT02538107
Title: Non-interventional, Observational Study to Investigate the Efficiency and Safety of Mircera in Patients With a Kidney Transplant
Brief Title: An Observational Study of Methoxy Polyethylene Glycol-epoetin Beta in Participants With a Kidney Transplant
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21386
Record Dates: First submitted 2015-08-24; First posted 2015-09-02 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Anemia, Kidney Transplantation
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Kidney Transplant Participants: Participants with kidney transplant and a chronic kidney disease who were receiving methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care.
  Interventions: Drug: Methoxy-polyethyleneglycol epoetin beta

INTERVENTIONS:
Drug: Methoxy-polyethyleneglycol epoetin beta
  Other Names: Mircera

SUMMARY:
This observational study will investigate efficacy and safety of methoxy polyethyleneglycol-epoetin beta in participants with a kidney transplant. Data of each participant will be collected over 15 months of Mircera therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with kidney transplant and a chronic kidney disease (CKD), who need erythropoiesis stimulating agent (ESA) therapy as part of their medical care and prescribed methoxy polyethyleneglycol-epoetin beta by the doctor.
* The transplant should function regularly and without need of continuous dialysis treatment at inclusion and also during the documentation period of this study according to treating physician's prognosis.

Exclusion Criteria:

* Kidney transplantation dates back less than 3 months. Acute decrease of hemoglobin (Hb) before enrollment, defined as decrease of greater than or equal to (>/=) 2 g/dL between two sequential values.
* Administration of other ESA therapies during the observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with kidney transplant prescribed methoxy polyethyleneglycol-epoetin beta
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2007-09-30 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2011-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Klinikum Hann. Münden, Nephrologisches Zentrum Niedersachsen, Hannoversch Münden, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Kidney Transplant Participants: Participants with chronic kidney disease who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
Period: Overall Study
Arm/Group | Kidney Transplant Participants
Started | 290
Completed | 180
Not Completed | 110
Not completed — Did not receive any Mircera dose | 11
Not completed — Missing | 5
Not completed — Necessity of dialysis | 20
Not completed — Administration of other ESA | 11
Not completed — No further treatment necessary | 18
Not completed — Withdrawal by Subject | 17
Not completed — Death | 4
Not completed — Administrative reason | 5
Not completed — Adverse Event | 4
Not completed — Surgery | 1
Not completed — Other | 7
Not completed — Not recorded | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants who received at least 1 dose of study treatment. Age was reported for N=278 participants since data for 1 participant was missing.
Arm/Group | Kidney Transplant Participants
Number analyzed (Participants) | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (14.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 142

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Hemoglobin Value of 11-12 Grams Per Deciliter (g/dL) From Visit 7 (Month 7) to Visit 9 (Month 9)
Time Frame: From Month 7 to Month 9
Population: Efficacy analysis set (Included participants who reported no pregnancy during the study period and had dosing and hemoglobin data available during 1 of the 3 visits [Visits 7-9]).
Measure: Number; unit: percentage of participants
Arm/Group | Kidney Transplant Participants
Number analyzed (Participants) | 193
percentage of participants | 20.7

2. Primary Outcome: Percentage of Participants With a Hemoglobin Value of 11-13 g/dL From Visit 7 (Month 7) to Visit 9 (Month 9)
Time Frame: From Month 7 to Month 9
Population: Efficacy analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Kidney Transplant Participants
Number analyzed (Participants) | 193
percentage of participants | 40.4

3. Primary Outcome: Percentage of Participants With a Hemoglobin Value of 11-13 g/dL From Visit 7 (Month 7) to Visit 12 (Month 12)
Time Frame: From Month 7 to Month 12
Population: Efficacy analysis set. Participants who were evaluable at the specified time frame were included.
Measure: Number; unit: percentage of participants
Arm/Group | Kidney Transplant Participants
Number analyzed (Participants) | 137
percentage of participants | 21.2

4. Primary Outcome: Percentage of Participants With a Hemoglobin Value of 11-13 g/dL From Visit 7 (Month 7) to Visit 15 (Month 15)
Time Frame: From Month 7 to Month 15
Population: Efficacy analysis set. Participants who were evaluable at the specified time frame were included.
Measure: Number; unit: percentage of participants
Arm/Group | Kidney Transplant Participants
Number analyzed (Participants) | 131
percentage of participants | 12.2

5. Primary Outcome: Percentage of Participants With a Hemoglobin Value of 10-13 g/dL From Visit 7 (Month 7) to Visit 12 (Month 12)
Time Frame: From Month 7 to Month 12
Population: Efficacy analysis set. Participants who were evaluable at the specified time frame were included.
Measure: Number; unit: percentage of participants
Arm/Group | Kidney Transplant Participants
Number analyzed (Participants) | 137
percentage of participants | 52.6

6. Secondary Outcome: Hemoglobin Level Based on the Type of Kidney Transplantation Performed
Description: Participants were classified based on the type of kidney transplantation they underwent before entering in to the study in to two groups; participants who received living donation and participants who received cadaveric donation.
Time Frame: Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 13, Month 14, Month 15 and Entire study (Month 1 to Month 15)
Population: Efficacy analysis set. n = number of participants who were evaluable at a particular visit.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Living Donation-Kidney Transplant Participants: Participants with chronic kidney disease who underwent 'living donation' type of kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
- Cadaveric Donation-Kidney Transplant Participants: Participants with chronic kidney disease who underwent 'cadaveric donation' type of kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
Arm/Group | Living Donation-Kidney Transplant Participants | Cadaveric Donation-Kidney Transplant Participants
Number analyzed (Participants) | 34 | 159
g/dL
  Visit 1 (Month 1) (n=22, 113) | 11.08 (1.244) | 11.26 (1.126)
  Visit 2 (Month 2) (n=25, 118) | 11.37 (1.215) | 11.41 (1.239)
  Visit 3 (Month 3) (n=27, 128) | 11.34 (1.163) | 11.71 (1.250)
  Visit 4 (Month 4) (n=23, 128) | 11.30 (1.213) | 11.56 (1.229)
  Visit 5 (Month 5) (n=25, 122) | 11.74 (1.174) | 11.75 (1.126)
  Visit 6 (Month 6) (n=20, 113) | 11.08 (0.896) | 11.66 (1.177)
  Visit 7 (Month 7) (n=21, 121) | 11.23 (1.132) | 11.59 (1.132)
  Visit 8 (Month 8) (n=24, 113) | 11.18 (1.305) | 11.57 (1.239)
  Visit 9 (Month 9) (n=17, 125) | 11.36 (1.386) | 11.60 (1.280)
  Visit 10 (Month 10) (n=21, 107) | 11.26 (1.435) | 11.59 (1.179)
  Visit 11 (Month 11) (n=18, 99) | 11.46 (1.079) | 11.62 (1.254)
  Visit 12 (Month 12) (n=22, 110) | 11.12 (1.437) | 11.41 (1.161)
  Visit 13 (Month 13) (n=23, 100) | 10.86 (1.386) | 11.32 (1.248)
  Visit 14 (Month 14) (n=18, 101) | 11.21 (1.018) | 11.35 (1.039)
  Visit 15 (Month 15) (n=21, 84) | 11.05 (1.187) | 11.50 (1.067)
  Entire study (Month 1 to Month 15) (n=34, 159) | 11.25 (0.853) | 11.49 (0.830)

7. Secondary Outcome: Hemoglobin Level Based on the Presence of Inflammatory Diseases
Description: Participants were classified based on the presence of other inflammatory diseases at baseline in to two groups; participants with presence of inflammatory diseases and participants with absence of inflammatory diseases.
Time Frame: as for outcome 6
Population: Efficacy analysis set. n = number of participants who were evaluable at a particular visit.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Inflammatory Diseases Present-Kidney Transplant Participants: Participants with chronic kidney disease and presence of other inflammatory diseases at baseline who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
- Inflammatory Diseases Absent-Kidney Transplant Participants: Participants with chronic kidney disease and absence of other inflammatory diseases at baseline who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
Arm/Group | Inflammatory Diseases Present-Kidney Transplant Participants | Inflammatory Diseases Absent-Kidney Transplant Participants
Number analyzed (Participants) | 56 | 137
g/dL
  Visit 1 (Month 1) (n=41, 94) | 11.30 (1.168) | 11.20 (1.137)
  Visit 2 (Month 2) (n=43, 100) | 11.33 (1.231) | 11.44 (1.236)
  Visit 3 (Month 3) (n=45, 110) | 11.75 (1.419) | 11.61 (1.163)
  Visit 4 (Month 4) (n=47, 104) | 11.54 (1.209) | 11.51 (1.240)
  Visit 5 (Month 5) (n=43, 104) | 11.71 (1.135) | 11.76 (1.133)
  Visit 6 (Month 6) (n=42, 91) | 11.34 (1.068) | 11.68 (1.184)
  Visit 7 (Month 7) (n=40, 102) | 11.46 (1.276) | 11.56 (1.080)
  Visit 8 (Month 8) (n=40, 97) | 11.58 (1.324) | 11.46 (1.230)
  Visit 9 (Month 9) (n=42, 100) | 11.61 (1.236) | 11.55 (1.318)
  Visit 10 (Month 10) (n=34, 94) | 11.63 (0.996) | 11.50 (1.300)
  Visit 11 (Month 11) (n=34, 83) | 11.75 (1.015) | 11.53 (1.302)
  Visit 12 (Month 12) (n=33, 99) | 11.23 (1.095) | 11.41 (1.248)
  Visit 13 (Month 13) (n=36, 87) | 11.17 (1.129) | 11.26 (1.346)
  Visit 14 (Month 14) (n=31, 88) | 11.07 (1.090) | 11.42 (1.003)
  Visit 15 (Month 15) (n=27, 78) | 11.03 (1.157) | 11.55 (1.056)
  Entire study (Month 1 to Month 15) (n=56, 137) | 11.38 (0.730) | 11.48 (0.878)

8. Secondary Outcome: Hemoglobin Level Based on the Etiology of Chronic Kidney Disease
Description: Participants were classified based on the etiology of chronic kidney disease. The different etiological reasons included diabetic vasculopathy, hypertensive nephrosclerosis, glomerulonephritis, polycystic kidney, chronic pyelonephritis, other reasons and origin unknown. Hemoglobin levels in participants who had etiology of chronic kidney disease as 'glomerulonephritis' or 'other reasons' were presented as these were the majority of the etiological reasons for chronic kidney disease.
Time Frame: as for outcome 6
Population: Efficacy analysis set. Participants who were evaluable for the specified group were included and n = number of participants who were evaluable at a particular visit.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Glomerulonephritis-Kidney Transplant Participants: Participants with glomerulonephritis as the cause of chronic kidney disease who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
- Other Reason-Kidney Transplant Participants: Participants with unspecified other reasons as the cause of chronic kidney disease who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
Arm/Group | Glomerulonephritis-Kidney Transplant Participants | Other Reason-Kidney Transplant Participants
Number analyzed (Participants) | 60 | 55
g/dL
  Visit 1 (Month 1) (n=43, 37) | 11.27 (1.254) | 11.44 (1.149)
  Visit 2 (Month 2) (n=43, 40) | 11.42 (1.240) | 11.48 (1.330)
  Visit 3 (Month 3) (n=49, 46) | 11.79 (1.298) | 11.75 (1.266)
  Visit 4 (Month 4) (n=49, 41) | 11.37 (1.270) | 11.76 (1.172)
  Visit 5 (Month 5) (n=46, 40) | 11.88 (1.156) | 11.72 (1.172)
  Visit 6 (Month 6) (n=40, 36) | 11.62 (1.129) | 11.68 (1.197)
  Visit 7 (Month 7) (n=46, 44) | 11.71 (1.270) | 11.52 (1.227)
  Visit 8 (Month 8) (n=39, 35) | 11.71 (1.305) | 11.60 (1.439)
  Visit 9 (Month 9) (n=45, 40) | 11.88 (1.126) | 11.46 (1.594)
  Visit 10 (Month 10) (n=44, 31) | 11.60 (1.266) | 11.67 (1.323)
  Visit 11 (Month 11) (n=33, 38) | 11.96 (1.236) | 11.47 (1.327)
  Visit 12 (Month 12) (n=36, 41) | 11.33 (1.452) | 11.37 (1.196)
  Visit 13 (Month 13) (n=41, 36) | 11.32 (1.530) | 11.20 (1.208)
  Visit 14 (Month 14) (n=40, 33) | 11.59 (1.077) | 11.26 (1.100)
  Visit 15 (Month 15) (n=35, 31) | 11.40 (1.296) | 11.47 (1.140)
  Entire study (Month 1 to Month 15) (n=60, 55) | 11.52 (0.924) | 11.52 (0.876)

9. Secondary Outcome: Hemoglobin Level Based on the Acute Bleeding Episode(s) During the Study
Description: Participants were classified in to two groups based on the presence of acute bleeding episodes during the study; presence or absence of bleeding episodes.
Time Frame: as for outcome 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Absence of Acute Bleeding-Kidney Transplant Participants: Participants with absence of acute bleeding episodes during the study with chronic kidney disease who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
- Presence of Acute Bleeding-Kidney Transplant Participants: Participants with presence of acute bleeding episodes during the study with chronic kidney disease who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
Arm/Group | Absence of Acute Bleeding-Kidney Transplant Participants | Presence of Acute Bleeding-Kidney Transplant Participants
Number analyzed (Participants) | 192 | 0
g/dL
  Visit 1 (Month 1) (n=135, 0) | 11.23 (1.143) |
  Visit 2 (Month 2) (n=142, 0) | 11.40 (1.231) |
  Visit 3 (Month 3) (n=155, 0) | 11.65 (1.240) |
  Visit 4 (Month 4) (n=150, 0) | 11.51 (1.229) |
  Visit 5 (Month 5) (n=147, 0) | 11.75 (1.130) |
  Visit 6 (Month 6) (n=132, 0) | 11.57 (1.159) |
  Visit 7 (Month 7) (n=141, 0) | 11.53 (1.139) |
  Visit 8 (Month 8) (n=137, 0) | 11.50 (1.254) |
  Visit 9 (Month 9) (n=141, 0) | 11.57 (1.294) |
  Visit 10 (Month 10) (n=128, 0) | 11.53 (1.224) |
  Visit 11 (Month 11) (n=116, 0) | 11.59 (1.231) |
  Visit 12 (Month 12) (n=132, 0) | 11.37 (1.210) |
  Visit 13 (Month 13) (n=122, 0) | 11.24 (1.285) |
  Visit 14 (Month 14) (n=118, 0) | 11.32 (1.035) |
  Visit 15 (Month 15) (n=104, 0) | 11.40 (1.101) |
  Entire study (Month 1 to Month 15) (n=192, 0) | 11.45 (0.839) |

10. Secondary Outcome: Hemoglobin Level Based on the Glomerular Filtration Rate (GFR)
Description: GFR is described as the flow rate of filtered fluid through the kidney and was determined using the Cockcroft-Gault formula to calculate the creatinine clearance. For males, creatinine clearance [milliliters per minute (mL/min)] = [(140 minus age) multiplied by (*) (body weight in kilogram [kg]) divided by [72 * serum creatinine milligrams per deciliter (mg/dL)]. For females, creatinine clearance (mL/min) = 0.85 * [(140 minus age) * (body weight in kg)] divided by [72 * serum creatinine (mg/dL)]. Participants were classified based on the GFR in to two groups; GFR less than (<) 30 mL/min and in the range of 30-60 mL/min and hemoglobin levels at different visits were presented.
Time Frame: as for outcome 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- GFR (<30 mL/Min)-Kidney Transplant Participants: Participants with GFR <30 mL/min with chronic kidney disease who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
- GFR (30-60 mL/Min)-Kidney Transplant Participants: Participants with GFR in the range of 30-60 mL/min with chronic kidney disease who underwent kidney transplantation and received methoxy polyethylene glycol epoetin beta (Mircera) as part of their medical care were observed and documented for up to 15 months.
Arm/Group | GFR (<30 mL/Min)-Kidney Transplant Participants | GFR (30-60 mL/Min)-Kidney Transplant Participants
Number analyzed (Participants) | 46 | 60
g/dL
  Visit 1 (Month 1) (n=35, 41) | 11.15 (0.952) | 11.44 (1.200)
  Visit 2 (Month 2) (n=35, 45) | 11.17 (1.234) | 11.42 (1.103)
  Visit 3 (Month 3) (n=40, 48) | 11.60 (1.205) | 11.65 (0.954)
  Visit 4 (Month 4) (n=37, 52) | 11.26 (1.242) | 11.75 (1.086)
  Visit 5 (Month 5) (n=37, 47) | 11.40 (1.090) | 11.87 (1.104)
  Visit 6 (Month 6) (n=34, 41) | 11.32 (1.158) | 11.90 (1.257)
  Visit 7 (Month 7) (n=36, 46) | 11.46 (1.108) | 11.62 (1.223)
  Visit 8 (Month 8) (n=28, 48) | 11.46 (1.215) | 11.66 (1.165)
  Visit 9 (Month 9) (n=38, 46) | 11.50 (1.369) | 11.85 (1.161)
  Visit 10 (Month 10) (n=30, 41) | 11.22 (1.063) | 11.88 (0.992)
  Visit 11 (Month 11) (n=30, 38) | 11.55 (1.071) | 11.69 (1.126)
  Visit 12 (Month 12) (n=27, 45) | 11.41 (0.943) | 11.67 (1.038)
  Visit 13 (Month 13) (n=31, 39) | 11.44 (1.048) | 11.41 (1.363)
  Visit 14 (Month 14) (n=27, 41) | 11.29 (1.056) | 11.40 (1.089)
  Visit 15 (Month 15) (n=24, 35) | 11.20 (1.093) | 11.81 (0.993)
  Entire study (Month 1 to Month 15) (n=46, 60) | 11.26 (0.784) | 11.62 (0.716)

11. Primary Outcome: Percentage of Participants With a Hemoglobin Value of 10-13 g/dL From Visit 7 (Month 7) to Visit 15 (Month 15)
Time Frame: From Month 7 to Month 15
Population: Efficacy analysis set. Participants who were evaluable at the specified time frame were included.
Measure: Number; unit: percentage of participants
Arm/Group | Kidney Transplant Participants
Number analyzed (Participants) | 131
percentage of participants | 41.2

12. Primary Outcome: Average Duration in Months Mircera Was Administered at Current Dose After the Previous Dose Adjustment
Time Frame: Up to 50 months
Population: Efficacy analysis set. Participants with non-missing values were included.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Kidney Transplant Participants
Number analyzed (Participants) | 192
months | 9.31 (6.250)

ADVERSE EVENTS:
Time Frame: Up to 50 months
Description: Safety analysis set.
Arm/Group | Kidney Transplant Participants
Serious Adverse Events (participants affected / at risk) | 32/279
Other Adverse Events (participants affected / at risk) | 42/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kidney Transplant Participants (N=279)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Device failure (General disorders) | 1
Inflammation (General disorders) | 1
Multi-organ failure (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Kidney transplant rejection (Immune system disorders) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis norovirus (Infections and infestations) | 1
Human polyomavirus infection (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Urinary tract infection enterococcal (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 4
C-reactive protein increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Weight decreased (Investigations) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
VIth nerve disorder (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Dialysis (Surgical and medical procedures) | 1
Haemodialysis (Surgical and medical procedures) | 1
Parathyroidectomy (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kidney Transplant Participants (N=279)
Bone marrow failure (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Macrocytosis (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Diplopia (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 4
Injection site pain (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 9
Oral herpes (Infections and infestations) | 3
Otitis media (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 6
Epicondylitis (Injury, poisoning and procedural complications) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Phantom pain (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1
Walking disability (Social circumstances) | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.